CLINICAL TRIAL: NCT00162526
Title: A Randomized Double Blind Placebo Controlled Clinical Trial Aim to Assess the Efficacy of Vitamin E Formulation (Tocopherol) in the Treatment of Chemotherapy Induced Stomatitis in Patients Undergoing Stem Cell Transplantation
Brief Title: Tocopherol is a Novel Treatment for Cancer Related Mucositis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the PI is no longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 270505-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2005-09

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Tocopherols

INTERVENTIONS:
Drug: Tocopherol

SUMMARY:
The present protocol is an attempt to prevent/treat mucositis in highly susceptible patients subjected to maximally tolerated doses of subsequently-myeloablative or myeloablative doses of chemoradiotherapy supported by autologous or allogeneic stem cell transplantation at the Department of Bone Marrow Transplantation. Mucositis is a major problem in the management of transplant recipients which subjects the patients to the risk of sepsis, need for parenteral nutrition and need of narcotics. We are planning a 2 arm study, comparing 2 safe vitamin E based formulations with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant and non-lactating females, 18 years of age or older at the time of screening, who are to receive myeloablative agonists with or without total body irradiation (TBI) in preparation for either allogeneic or autologous HSCT. Patients who are to be hospitalized and are expected to remain hospitalized until marrow recovery.
* Karnofsky performance status of 60 or greater or ECOG performance status of 2 or less.
* Normal dental examination as assessed by the investigator.

Exclusion Criteria:

* Clinically significant acute and active oral cavity infection.
* Patients taking any investigational or other non-approved oral therapy for oral mucositis.
* Known hypersensitivity to Vitamin E.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-12

PRIMARY OUTCOMES:
To evaluate the tolerability and the safety of a Tocopherol formulation in the prevention or suppression of the serverity of oral mucositis induced by myeloablative agonist.

SECONDARY OUTCOMES:
To evaluate the toxicity and the safety of a Tocopherol formulation in the prevention or suppression of the serverity of oral mucositis induced by myeloablative agonist.

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel